CLINICAL TRIAL: NCT01463553
Title: Improving Primary Spontaneous Pneumothorax (PSP) Treatment Techniques in VATS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Haidian Hospital (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Huang Yuqing, Deputy Director, Beijing Haidian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z111107058811089
Record Dates: First submitted 2011-10-30; First posted 2011-11-02 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Pneumothorax; Pleurodesis
Keywords: primary spontaneous pneumothorax; VATS; pleurodesis; recurrence rate
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wedge resection (No Intervention)
- Wedge resection and pleurodosis (Experimental)
  Interventions: Procedure: VATS pleurodesis

INTERVENTIONS:
Procedure: VATS pleurodesis — Based on the findings, establish selection standards for the timing of surgery to treat PSP by VATS and establish technical specifications for performing operations on different types of lung bullae. The goal is to improve the diagnosis and treatment of PSP so as to reduce the recurrence rate of pneumothorax, reduce the trauma of operation, shorten hospital stays and postoperative recovery time, and provide better services for returning to everyday life and improving the quality of life for patients.
  Arms: Wedge resection and pleurodosis

SUMMARY:
The purpose of this study is to:

1. Evaluate the validity of using abnormal characteristics of the pneumothorax line, as evaluated from chest X-ray film, as the operative indications for video-assisted thoracic surgery (VATS) on primary spontaneous pneumothorax (PSP).
2. Through a randomized double blind controlled trial on patients whose PSP was caused by lung bullae, evaluate the effectiveness of pleurodesis in terms of the rate of recurrence of PSP and the trauma of the operation on patients.
3. Based on the findings, establish selection standards for the timing of surgery to treat PSP by VATS and establish technical specifications for performing operations on different types of lung bullae. The goal is to improve the diagnosis and treatment of PSP so as to reduce the recurrence rate of pneumothorax, reduce the trauma of operation, shorten hospital stays and postoperative recovery time, and provide better services for returning to everyday life and improving the quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients in whom obvious bullous forms are seen in PSP pneumothorax lines, or whose pneumothorax lines are rough and interrupted with or without thoracentesis, thoracic close drainage
2. patients whose lung compression exceeded 30% for the first incidence of pneumothorax
3. patients between the ages of 14 and 40, with normal vital signs (body temperature, breathing, blood pressure, pulse) and normal results on routine examination (routine blood test, liver and kidney functions)
4. no language barrier, such as surdimutism, aphasia
5. patients who voluntarily joined the group and signed the informed consent after reviewing the substance, significance and risks of this experiment

Exclusion Criteria:

1. patients who refuse VATS operation
2. patients who refuse the follow-up
3. patients with secondary spontaneous pneumothorax including that caused by emphysema, COPD, asthma, pulmonary lymphangiomyomatosis, thoracic injury and other diseases
4. patients with mental illness, low IQ, or inability to understand the informed consent
5. substance abusers

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Primary Spontaneous Pneumothorax (PSP) | 24 months
  Monitor patients for 24 months to measure recurrence rate of primary spontaneous pneumothorax

SECONDARY OUTCOMES:
Did not recurrence | 24months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, associate director, Principal Investigator — Peking University People Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Min X, Huang Y, Yang Y, Chen Y, Cui J, Wang C, Huang Y, Liu J, Wang J. Mechanical pleurodesis does not reduce recurrence of spontaneous pneumothorax: a randomized trial. Ann Thorac Surg. 2014 Nov;98(5):1790-6; discussion 1796. doi: 10.1016/j.athoracsur.2014.06.034. Epub 2014 Sep 16. PMID 25236367